CLINICAL TRIAL: NCT02876354
Title: Risk Factors for Vascular Calcifications in Hemodialysis Patients: to What Extent is Vitamin K2 Deficiency Involved?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Mabel Aoun, Head of the Department of Nephrology, Saint-Georges Hospital Ajaltoun, Saint-Joseph University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGH001
Record Dates: First submitted 2016-08-11; First posted 2016-08-23 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Vascular Calcifications
Keywords: Hemodialysis; Vitamin k2; Vascular calcifications
MeSH Terms: conditions — Vascular Calcification | interventions — Vitamin K 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Menaquinone 360 (Experimental): All patients in the study will be assigned to receive menaquinone 360 μg /d for 4 weeks.
  Interventions: Drug: Menaquinone

INTERVENTIONS:
Drug: Menaquinone — Patients on hemodialysis will be supplemented by 360 μg /d of menaquinone for 4 weeks. At baseline they will have a lateral abdominal X-Ray and dosage of dp-ucMGP. At the end of the study patients will have a second measurement of dp-ucMGP levels.
  Other Names: Vitamin k2

SUMMARY:
Vitamin K2 deficiency has been shown to be profound in hemodialysis patients. It is reflected by high plasma levels of dephosphorylated-undercarboxylated Matrix Gla protein (dp-ucMGP) and seems to be correlated with vascular calcifications. Vascular calcifications can be assessed using the AC24 score on a lateral abdominal X-ray.

The aim of this study is to assess first the rate of decrease of dp-ucMGP in a hemodialysis cohort after supplementation with vitamin K2 and the correlation between this rate of decrease and the Aortic Calcification Severity (AC24) score. The factors associated with high levels of dp-ucMGP will be analyzed as well.

DETAILED DESCRIPTION:
Background The majority of patients reaching end-stage renal disease (ESRD) and dialysis have vascular calcifications. Those vascular calcifications tend to increase mortality in this specific population. It has been shown that high scores of vascular calcifications in a healthy patient with no cardiovascular risk factors lead to a higher mortality rate compared with someone with ≥3 risk factors without calcification. In hemodialysis (HD) patients, cardiovascular risk factors are numerous and they include the traditional ones such as age, smoking, diabetes, hypertension, hyperlipidemia and those specific to chronic kidney disease (CKD) as for instance hyperparathyroidism. All those facts are compelling arguments to look seriously for a treatment against vascular calcifications. Therefore the 2009 Kidney disease: Improving Global Outcomes (KDIGO) Clinical Practice Guideline for the Diagnosis, Evaluation, Prevention, and Treatment of Chronic Kidney Disease-Mineral and Bone Disorder (CKD-MBD) has suggested to measure those vascular calcifications scores by a lateral abdominal radiograph that is a cost-effective alternative to the standard computed tomography-based imaging.

In order to lower or prevent vascular calcifications in chronic kidney disease (CKD) patients, many interventions have been studied in the past. They have included treatments such as statins, non-calcium-based phosphate binders and cinacalcet. So far, the non-calcium-based phosphate binders showed significant benefit on mortality but none of the studies manifested a solid beneficial effect on vascular calcifications.

In the last years, remarkable data emerged concerning the association between vascular calcifications and plasmatic levels of dephosphorylated-undercarboxylated MGP (dp-ucMGP). dp-ucMGP is the inactive form of Matrix gla protein (MGP). MGP is a small protein known to act locally in the tissues as a calcification inhibitor and it is vitamin K dependent. High dp-ucMGP levels reflect low activity of MGP. Vitamin K2 deficiency is one of the factors that increase dp-ucMGP. There have been several reports also showing that dp-ucMGP levels increase gradually after the age of 40 and are significantly higher in those older than 65, in patients with diabetes, aortic stenosis, heart failure and on vitamin K antagonists (VKA). They are also extremely high in ESRD patients on dialysis. Moreover the combination of VKA and dialysis increases the incidence of calciphylaxis.

Since high dp-ucMGP levels suggest vitamin k2 deficiency and are associated with vascular calcification, supplementing high-risk patients especially CKD patients with vitamin k2 (menaquinone) seems very promising. Vitamin k2 can be provided to the patient as a pill or through a specific food diet. Food that seems to affect dp-ucMGP levels includes natto and fermented cheese such as camembert, goat cheese or gouda.

Vitamin K2 supplementation was analyzed in several European HD cohorts. In 2012, Westenfeld et al. demonstrated that vitamin k2 supplements in hemodialysis patients lead to a dose-dependent decrease in plasma dp-ucMGP levels. This was reproduced by Caluwé at al in 2014 and they both showed that a dose of 360 μg /d lower the dp-ucMGP by 30-33%.

Studies in patients with normal renal function showed a higher decrease of dp-ucMGP ~50% under 180 μg /d of menaquinone and this could be explained in many ways. Either vitamin K2 deficiency is very profound in CKD and particularly dialysis patients or dp-ucMGP does not only reflect vitamin k2 deficiency in those patients. High dp-ucMGP could be associated with other risk factors for calcifications in chronic kidney disease such as phosphate, calcium or parathyroid hormone (PTH).

Middle-Eastern diet is different from European countries and MGP activity as well as vitamin K2 supplementation have not yet been studied in dialysis populations in this part of the world.

Therefore this study will be conducted in a Lebanese hemodialysis center where patients will receive vitamin k2 for 4 weeks. The investigators will assess first the rate of decrease of dp-ucMGP after supplementation with vitamin K2 and the correlation between this rate of decrease and the AC24 score. They will analyze as well the factors associated with high levels of dp-ucMGP. Finally they will define the rate of decrease of dp-ucMGP after VKA withdrawal in a small subgroup before including them in the study.

Methods and design

Trial design, participants and data collection This is a prospective, pre-post intervention clinical trial. All patients in a single dialysis center older than 18 years on chronic hemodialysis since more than one month will be included. Patients who are taking VKA and can not stop it (heart valve replacement cases) will be excluded. The total expected trial duration is 4 weeks.

Data for demographics, comorbidities, medications and laboratory results are collected from the patients' medical records. Variables that will be studied are: age, gender, months on dialysis, residual diuresis, BMI, urea reduction ratio (URR), diabetes, hypertension, smoking, hyperlipidemia, calcium and non-calcium-based phosphate binders, cinacalcet, alfacalcidol, AC-24 score, dp-ucMGP level, albumin, coronary artery disease, mean of calcium, phosphorus and parathyroid hormone (PTH).

Calcium, phosphorus, PTH, LDL cholesterol and serum albumin levels will be collected from the medical record of the patient. Calcium and phosphorus are measured monthly on a routine basis; the mean of the last 12 measurements will be calculated. PTH is measured every 4-6 months; all PTH levels of each patient will be collected since the start of dialysis in order to obtain the mean PTH level.

Definitions Coronary artery disease is defined as a history of coronary artery disease treated medically or interventionally. Diabetes and hypertension are defined as taking antidiabetic treatment or antihypertensive treatment respectively.

Normal phosphate and calcium are defined respectively as 3.5-4.5 mg/dL and 8.4-9.5 mg/dL.

Non-calcium phosphate binders available are sevelamer and lanthanum. The only active vitamin D that patients will take is alfacalcidol.

Ethical considerations The study is approved by the ethical committee of the Saint-Joseph University-Beirut and complies with the Declaration of Helsinki of 1975. All patients have to give written informed consent to participate.

The supplementation with vitamin K2 does not put the patient at risk of hypercoagulability and a previous prospective cohort of 35000 healthy subjects supplemented with vitamin K showed no increase in ischemic stroke events.

Intervention:

Patients will be eligible for the trial if they sign the informed consent. All patients will receive 360 μg of menaquinone once daily. Menaquinone will be provided by Omicron, Lebanon. The chosen dose in this trial was established from two previous trials done on hemodialysis patients. A daily dose of 360 μg Menaquinone reduces the amount of inactive MGP by 30-33% in hemodialysis patients. The dose of the day of dialysis will be given in the center to ensure at least the compliance towards the half of the dose per week.

Before starting the trial, patients on vitamin k antagonists as a prevention for vascular access thrombosis will withdraw the VKA and be included in the study after stabilization of their dp-ucMGP levels. The investigators will assess the average time necessary to reach a stable level of dp-ucMGP after VKA withdrawal. Patients will be assigned to receive 360 μg of menaquinone once daily.

Analysis of dp-ucMGP and AC-24 score measurements dp-ucMGP will be measured twice, once before the vitamin k2 supplementation and second after four weeks of the treatment. Pre-dialysis venous blood samples will be processed to the same laboratory.

Circulating dp-ucMGP will be quantified using a dual antibody enzyme-linked immunosorbent assay provided by Immunodiagnostic Systems Ltd, United Kingdom.

Lateral abdominal X-ray of the lumbar aorta will be performed at the inclusion of the study. For each patient the abdominal aortic calcifications will be estimated using the Aortic Calcification Severity (AC-24) score. The AC-24 score will be calculated by two independent physicians. If the difference is one point, the higher score will be recorded. If the difference is more than one point a third opinion will be sought and the mean of the three levels will be retained.

Clinical data and Follow-up Patients will have their pre-dialysis blood pressure measured after 15 min of rest and recorded at the beginning and the end of the study using validated automated electronic monitors. Their blood pressure levels will be checked also during the 4 weeks period three times per week in the dialysis center.

Assessment of adverse events Patients will be evaluated for any side-effect at each dialysis session, especially regarding their vascular access patency or other thrombotic event.

Statistical analysis Descriptive statistics will be used to represent important variables of known risk factors, exposures and treatment options. Continuous variables that are normally distributed will be presented as means and standard deviation. Otherwise median and range will be the appropriate method. Student t test and one way ANOVA will be used for parametric variables comparison and Mann Whitney U and Kruskal Wallis for non parametric variables. Categorical variables will be presented by count and percentage. Χ2 fischer exact test and logistic regression will be used to compare two or more categorical variables respectively.

Pearson correlation will be calculated to investigate the association of vascular calcifications score with dp-ucMGP level as well as with potential covariates. A stepwise multivariable linear regression will be employed to adjust for the association of MGP with calcification score in the presence of significant covariates. P < 0.20 will be considered valid for inclusion in the model. A 2-sided P < 0.05 will be considered significant. To determine the effect of vitamin K2 intake on dp-ucMGP, the pre- and post-levels will be compared using matched t-test. All analyses will be done using SPSS statistics (22.0 version, SPSS Inc, Chicago, III).

ELIGIBILITY:
Inclusion Criteria:

* Patients on chronic hemodialysis in our center older than 18 years old who sign the informed consent.

Exclusion Criteria:

* Patients who are not eligible for a discontinuation of vitamin k antagonists

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Rate of decrease of dp-ucMGP after daily supplementation with menaquinone | Baseline-Four weeks
  We will analyze whether the percentage of decrease of dp-ucMGP in our Middle-Eastern country following vitamin k2 supplementation is similar to that reported in the previous trials in Europe.

CONTACTS AND LOCATIONS:
Overall Officials: Mabel Aoun, MD, Principal Investigator — Université Saint-Joseph, Beirut, Lebanon
Locations (1):
- Saint-Georges Hospital, Ajaltoun, Keserwan, Lebanon

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Aoun M, Makki M, Azar H, Matta H, Chelala DN. High Dephosphorylated-Uncarboxylated MGP in Hemodialysis patients: risk factors and response to vitamin K2, A pre-post intervention clinical trial. BMC Nephrol. 2017 Jun 7;18(1):191. doi: 10.1186/s12882-017-0609-3. PMID 28592319